CLINICAL TRIAL: NCT04999111
Title: A Randomized, Double-blind, Phase 2 Study to Evaluate the Immunogenicity, Reactogenicity and Safety of Ad26.COV2.S Administered as Booster Vaccination in Adults 18 Years of Age and Older Who Have Previously Received Primary Vaccination With Ad26.COV2.S or BNT162b2
Brief Title: A Study of Ad26.COV2.S Administered as Booster Vaccination in Adults Who Have Previously Received Primary Vaccination With Ad26.COV2.S or BNT162b2
Acronym: Amplify
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR109060; VAC31518COV2008 (Other: Janssen Vaccines & Prevention B.V.)
Expanded Access: NCT04817657 (No longer available)
Record Dates: First submitted 2021-08-03; First posted 2021-08-10 (Actual); Results first posted 2023-01-05 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Coronavirus Disease
MeSH Terms: interventions — Ad26COVS1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: Group 1: Ad26.COV2.S (Dose Level 1) (Experimental): Participants who have previously received primary vaccination with Ad26.COV2.S will receive single intramuscular (IM) injection of Ad26.COV2.S booster vaccination at dose level 1 on Day 1.
  Interventions: Biological: Ad26.COV2.S
- Cohort 1: Group 2: Ad26.COV2.S (Dose Level 2) (Experimental): Participants who have previously received primary vaccination with Ad26.COV2.S will receive single IM injection of Ad26.COV2.S booster vaccination at dose level 2 on Day 1.
  Interventions: Biological: Ad26.COV2.S
- Cohort 1: Group 3: Ad26.COV2.S (Dose Level 3) (Experimental): Participants who have previously received primary vaccination with Ad26.COV2.S will receive single IM injection of Ad26.COV2.S booster vaccination at dose level 3 on Day 1.
  Interventions: Biological: Ad26.COV2.S
- Cohort 2: Group 4: Ad26.COV2.S (Dose Level 1) (Experimental): Participants who have previously received primary vaccination with BNT162b2 will receive single IM injection of Ad26.COV2.S booster vaccination at dose level 1 on Day 1.
  Interventions: Biological: Ad26.COV2.S
- Cohort 2: Group 5: Ad26.COV2.S (Dose Level 2) (Experimental): Participants who have previously received primary vaccination with BNT162b2 will receive single IM injection of Ad26.COV2.S booster vaccination at dose level 2 on Day 1.
  Interventions: Biological: Ad26.COV2.S
- Cohort 2: Group 6: Ad26.COV2.S (Dose Level 3) (Experimental): Participants who have previously received primary vaccination with BNT162b2 will receive single IM injection of Ad26.COV2.S booster vaccination at dose level 3 on Day 1.
  Interventions: Biological: Ad26.COV2.S

INTERVENTIONS:
Biological: Ad26.COV2.S — Participants will receive IM injection of Ad26.COV2.S.
  Other Names: JNJ-78436735; VAC31518

SUMMARY:
The purposes of this study are to demonstrate the non-inferiority (NI) of the neutralizing antibody response to the original strain 14 days after booster vaccination with Ad26.COV2.S at the different dose levels, administered greater than or equal to (>=) 6 months after single-dose primary vaccination with Ad26.COV2.S, compared to the neutralizing antibody response to the original strain induced by single-dose primary vaccination with Ad26.COV2.S; To demonstrate the NI of the neutralizing antibody response to the leading variant of high consequence or concern 14 days after booster vaccination with Ad26.COV2.S at the 5*10^10 virus particle (vp) dose level, administered >= 6 months after single-dose primary vaccination with Ad26.COV2.S (5*10^10 vp dose level), compared to the neutralizing antibody response to the leading variant of high consequence or concern induced by single-dose primary vaccination with Ad26.COV2.S at the 5*10^10 vp dose level, if feasible; To demonstrate the NI of the neutralizing antibody response to the original strain 14 days after booster vaccination with Ad26.COV2.S at the different dose levels administered >=6 months after completing a 2-dose primary vaccination with Pfizer BNT162b2, compared to the neutralizing antibody response to the original strain induced by 2-dose primary vaccination with Pfizer BNT162b2; To demonstrate the NI of neutralizing antibody response to the leading variant of high consequence or concern 14 days after booster vaccination with Ad26.COV2.S at the 5*10^10 vp dose level, administered >= 6 months after completing a 2-dose primary vaccination with Pfizer BNT162b2, compared to the neutralizing antibody response to the leading variant of high consequence or concern induced by 2-dose primary vaccination with Pfizer BNT162b2, if feasible.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Participant received Ad26.COV2.S in VAC31518COV3001. The interval between the Ad26.COV2.S primary vaccination should preferably be greater than or equal to (>=) 6 months prior to study vaccination on VAC31518COV2008, however a window of maximum -20 days is allowed; Cohort 2: Participant completed primary vaccination with a 2-dose regimen of BNT162b2 vaccine. The last dose of BTN162b2 should preferably be >=6 months prior to study vaccination on COV2008, however a window of a maximum of -20 days is allowed
* Participant must provide consent indicating that he or she understands the purpose, procedures and potential risks and benefits of the study, and is willing to participate in the study
* Participant agrees to not donate bone marrow, blood, and blood products from the study vaccine administration until 3 months after receiving the study vaccine
* Participant must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study
* Participant must be able to read, understand, and complete questionnaires in the electronic clinical outcome assessment (eCOA) (that is, the Coronavirus disease (COVID-19) signs and symptoms surveillance question, the e-Diary, and the electronic patient-reported outcomes (ePROs). Participants with visual impairment are eligible for study participation and may have caregiver assistance in completing the eCOA questionnaires

Exclusion Criteria:

* Participant has a clinically significant acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature >= 38.0 degree Celsius (C) (100.4 degree Fahrenheit [F]) within 24 hours prior to the planned study vaccination; randomization at a later date is permitted at the discretion of the investigator. Please notify the sponsor (or medical monitor) of this decision
* Participant has a known or suspected allergy or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients (including specifically the excipients of the study vaccine
* Participant received treatment with immunoglobulins (Ig) in the 3 months or exogenous blood products (autologous blood transfusions are not exclusionary) in the 4 months before the planned administration of the study vaccine or has any plans to receive such treatment during the study
* Participant has a known history of confirmed severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) infection
* Participant has a history of heparin-induced thrombocytopenia or thrombosis in combination with thrombocytopenia
* Participant has a history of acute polyneuropathy (example. Guillain-Barre syndrome)
* History of capillary leak syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1541 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2022-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (21):
- United States (21):
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Synexus Clinical Research US Inc, Tucson, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Ark Clinical Research, Long Beach, California
  - Velocity Clinical Research, North Hollywood, California
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Research Centers of America, LLC, Hollywood, Florida
  - Synexus Clinical Research US Inc, Orlando, Florida
  - Synexus Clinical Research US Inc, The Villages, Florida
  - Optimal Research, Peoria, Illinois
  - Johnson County Clin-Trials, Lenexa, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Center for Virology and Vaccine Research, Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Rochester Clinical Research, Inc, Rochester, New York
  - Velocity Clinical Research, Anderson, Anderson, South Carolina
  - Accellacare US Inc, Mt. Pleasant, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Crofoot Research Center, Houston, Texas
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Roels S, Bruckner M, Sadoff J, Cardenas V, Tang C, Hagedoorn S, Heerwegh D, Stieh DJ, Le Gars M. Pre- and post-Ad26.COV2.S booster dose antibody levels predict COVID-19 disease risk. Vaccine. 2024 Sep 17;42(22):126159. doi: 10.1016/j.vaccine.2024.126159. Epub 2024 Aug 8. PMID 39121698
- [Derived] Le Gars M, Sadoff J, Cardenas V, Heerwegh D, Tesfaye F, Roey GV, Spicer C, Matias SS, Crayne O, Kamphuis T, Struyf F, Schuitemaker H, Douoguih M. Safety, reactogenicity, and immunogenicity of Ad26.COV2.S as homologous or heterologous COVID-19 booster vaccination: Results of a randomized, double-blind, phase 2 trial. Vaccine. 2024 Jul 25;42(19):3938-3952. doi: 10.1016/j.vaccine.2024.03.079. Epub 2024 Jun 25. PMID 38918103

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who received primary vaccination with Ad26.COV2.S and BNT162b2 were enrolled in this study. 1541 participants were enrolled in the study, of which 1532 participants were randomized in the study and vaccinated.
Groups:
- Cohort 1: Ad26.COV2.S (5*10^10 vp): Participants who had received primary vaccination with Ad26.COV2.S (1 dose) in study VAC31518COV3001 (NCT04505722) were enrolled in this study and received a single intramuscular (IM) injection of Ad26.COV2.S booster vaccination at 5*10^10 virus particle (vp) dose level on Day 1.
- Cohort 1: Ad26.COV2.S (2.5*10^10 vp): Participants who had received primary vaccination with Ad26.COV2.S (1 dose) in study VAC31518COV3001 (NCT04505722) were enrolled in this study and received a single IM injection of Ad26.COV2.S booster vaccination at 2.5*10^10 vp dose level on Day 1.
- Cohort 1: Ad26.COV2.S (1*10^10 vp): Participants who had received primary vaccination with Ad26.COV2.S (1 dose) in study VAC31518COV3001 (NCT04505722) were enrolled in this study and received a single IM injection of Ad26.COV2.S booster vaccination at 1*10^10 vp dose level on Day 1.
- Cohort 2: Ad26.COV2.S (5*10^10 vp): Participants who had received primary vaccination with BNT162b2 (2 doses) were enrolled in this study and received a single IM injection of Ad26.COV2.S booster vaccination at 5*10^10 vp dose level on Day 1.
- Cohort 2: Ad26.COV2.S (2.5*10^10 vp): Participants who had received primary vaccination with BNT162b2 (2 doses) were enrolled in this study and received a single IM injection of Ad26.COV2.S booster vaccination at 2.5*10^10 vp dose level on Day 1.
- Cohort 2: Ad26.COV2.S (1*10^10 vp): Participants who had received primary vaccination with BNT162b2 (2 doses) were enrolled in this study and received a single IM injection of Ad26.COV2.S booster vaccination at 1*10^10 vp dose level on Day 1.
Period: Overall Study
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp) | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Started (Enrolled Participants) | 331 | 328 | 116 | 329 | 331 | 106
Randomized and Vaccinated | 330 | 326 | 116 | 326 | 328 | 106
Completed | 277 | 271 | 96 | 260 | 251 | 84
Not Completed | 54 | 57 | 20 | 69 | 80 | 22
Not completed — Lost to Follow-up | 21 | 16 | 2 | 26 | 30 | 6
Not completed — Physician Decision | 1 | 3 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 23 | 29 | 15 | 30 | 35 | 10
Not completed — Other | 6 | 6 | 3 | 8 | 8 | 5
Not completed — Non-compliance with study schedule | 1 | 0 | 0 | 1 | 1 | 1
Not completed — Randomized but not vaccinated | 1 | 2 | 0 | 3 | 3 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Initiated prohibited medication | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants with a documented study vaccine administration (Ad26.COV2.S).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp) | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp) | Total
Number analyzed (Participants) | 330 | 326 | 116 | 326 | 328 | 106 | 1532
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (14.84) | 56.4 (13.88) | 56.2 (13.52) | 47.2 (15.38) | 47.9 (15.12) | 50 (17.98) | 51.9 (15.5)
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 234 | 226 | 84 | 275 | 268 | 75 | 1162
  From 65 to 84 years | 94 | 99 | 31 | 51 | 59 | 31 | 365
  85 years and over | 2 | 1 | 1 | 0 | 1 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 155 | 58 | 190 | 185 | 68 | 815
  Male | 171 | 171 | 58 | 136 | 143 | 38 | 717
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 46 | 15 | 38 | 38 | 8 | 183
  Not Hispanic or Latino | 274 | 264 | 101 | 281 | 281 | 97 | 1298
  Unknown or Not Reported | 18 | 16 | 0 | 7 | 9 | 1 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 0 | 0 | 1 | 0 | 6
  Asian | 15 | 11 | 6 | 12 | 19 | 5 | 68
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 1 | 4 | 0 | 7
  Black or African American | 32 | 25 | 4 | 12 | 20 | 9 | 102
  White | 275 | 275 | 103 | 292 | 279 | 91 | 1315
  More than one race | 3 | 6 | 1 | 3 | 3 | 0 | 16
  Unknown or Not Reported | 4 | 4 | 1 | 6 | 2 | 1 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 330 | 326 | 116 | 326 | 328 | 106 | 1532

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Percentage of Participants With Serological Response Against SARS-CoV-2 Original Strain 14 Days After Ad26.COV2.S Booster Vaccination After Completing Primary Vaccination With Ad26.COV2.S
Description: Percentage of participants with serological response against SARS-CoV-2 original strain (Wuhan, 2019, whole genome sequence) 14 days after Ad26.COV2.S booster vaccination after completing primary vaccination with Ad26.COV2.S was reported. A participant was considered a responder if one or both of the following conditions were satisfied: (1) Pre-booster titer less than (<) lower limit of quantification (LLOQ) and post-booster titer greater than or equal to (>=) 4*LLOQ or (2) Pre-booster titer greater than (>) LLOQ and post-booster titer >=4*pre-booster titer value.
Time Frame: 14 days after Ad26.COV2.S booster vaccination (i.e., on Day 15)
Population: Non-inferiority (NI) analysis set included all vaccinated participants with post-baseline immunogenicity data without major protocol deviations and who were SARS-COV-2 seronegative at baseline (based on the serological test for SARS CoV-2-specific nucleocapsid antibodies [N serology]). Here, N (Overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 298 | 297 | 93
Percentage of participants | 63.4 [57.7 to 68.9] | 57.9 [52.1 to 63.6] | 64.5 [53.9 to 74.2]

2. Primary Outcome: Cohort 1: Geometric Mean Titers (GMTs) of Neutralizing Antibodies Against SARS-CoV-2 Original Strain 14 Days After Ad26.COV2.S Booster Vaccination After Completing Primary Vaccination With Ad26.COV2.S
Description: GMTs of neutralizing antibodies against SARS-CoV-2 original strain 14 days after Ad26.COV2.S booster vaccination after completing primary vaccination with Ad26.COV2.S (5×10^10 vp dose level) were reported. GMT against original strain was assessed by virus neutralization assay (VNA).
Time Frame: 14 days after Ad26.COV2.S booster vaccination (i.e., on Day 15)
Population: NI analysis set included all vaccinated participants with post-baseline immunogenicity data without major protocol deviations and who were SARS-COV-2 seronegative at baseline (based on the serological test for SARS CoV-2-specific nucleocapsid antibodies [N serology]). Here, N (overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 298 | 297 | 93
Titer | 1130 [989 to 1291] | 915 [792 to 1058] | 734 [564 to 954]

3. Primary Outcome: Cohort 1: Percentage of Participants With Serological Response Against SARS-CoV-2 Original Strain 28 Days After Primary Vaccination With Ad26.COV2.S
Description: Percentage of participants with serological response against SARS-CoV-2 original strain 28 days after primary vaccination with Ad26.COV2.S (5×10^10 vp dose level) were reported. A participant was considered a responder if one or both of the following conditions were satisfied: (1) Pre-dose titer <LLOQ and post-vaccination titer >=4*LLOQ or (2) Pre-dose titer >LLOQ and post-vaccination titer >=4*pre-dose 1 titer value.
Time Frame: 28 days after primary vaccination with Ad26.COV2.S (Day 29 of study VAC31518COV3001)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 312 | 315 | 111
Percentage of participants | 15.4 [11.6 to 19.9] | 16.8 [12.9 to 21.4] | 11.7 [6.4 to 19.2]

4. Primary Outcome: Cohort 1: GMTs of Neutralizing Antibodies Against SARS-CoV-2 Original Strain 28 Days After Primary Vaccination With Ad26.COV2.S
Description: GMTs of neutralizing antibodies against SARS-CoV-2 original strain 28 days after primary vaccination with Ad26.COV2.S (5×10^10 vp dose level) were reported. GMT against original strain was assessed by VNA.
Time Frame: 28 days after primary vaccination with Ad26.COV2.S (Day 29 of study VAC31518COV3001)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 312 | 315 | 112
Titer | 98 [85 to 113] | 100 [87 to 115] | 76 [NA to 92] — Lower limit of 95% CI could not be estimated as it was below the LLOQ (75).

5. Primary Outcome: Cohort 1: Percentage of Participants With Serological Response Against the Delta Variant 14 Days After Ad26.COV2.S Booster Vaccination (5*10^10 vp Dose Level) After Completing Primary Vaccination With Ad26.COV2.S
Description: Percentage of participants with serological response against leading variant of high consequence or concern (delta variant) 14 days after Ad26.COV2.S booster vaccination (5*10^10 vp Dose Level) after completing primary vaccination with Ad26.COV2.S were reported. A participant was considered a responder if one or both of the following conditions were satisfied: (1) Pre-booster titer <LLOQ and post-booster titer >=4*LLOQ or (2) Pre-booster titer >LLOQ and post-booster titer >=4*pre-booster titer value. As specified in the protocol, data for this outcome measure was not collected and analyzed for Cohort 1: Ad26.COV2.S 2.5*10^10 vp and 1*10^10 vp participants.
Time Frame: 14 days after Ad26.COV2.S booster vaccination (i.e., On Day 15)
Population: NI analysis set included all vaccinated participants with post-baseline immunogenicity data without major protocol deviations and who SARS-COV-2 seronegative at baseline (based on the serological test for SARS CoV-2-specific nucleocapsid antibodies [N serology]). Here, N (Overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp)
Number analyzed (Participants) | 298
Percentage of participants | 56.7 [50.9 to 62.4]

6. Primary Outcome: Cohort 1: GMTs of Neutralizing Antibodies Against the Leading Variant of High Consequence or Concern (Delta Variant) 14 Days After Ad26.COV2.S Booster Vaccination (5*10^10 vp Dose Level) After Completing Primary Vaccination With Ad26.COV2.S
Description: GMTs of neutralizing antibodies against leading variant of high consequence or concern (delta variant) 14 days After Ad26.COV2.S booster vaccination (5*10^10 vp dose level) after completing primary vaccination with Ad26.COV2.S were reported. GMT against Delta Variant was assessed by VNA. As specified in the protocol, data for this outcome measure was not collected and analyzed for Cohort 1: Ad26.COV2.S 2.5*10^10 vp and 1*10^10 vp participants.
Time Frame: 14 days after Ad26.COV2.S booster vaccination (i.e., On Day 15)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp)
Number analyzed (Participants) | 298
Titer | 471 [411 to 539]

7. Primary Outcome: Cohort 1: Percentage of Participants With Serological Response Against SARS-CoV-2 Leading Variant of High Consequence or Concern (Delta Variant) 28 Days After Primary Vaccination With Ad26.COV2.S
Description: Percentage of participants with serological response against SARS-CoV-2 leading variant of high consequence or concern (delta variant) 28 days after primary vaccination with Ad26.COV2.S (5*10^10 vp dose level) were reported. A participant was considered a responder if one or both of the following conditions were satisfied: (1) Pre-dose titer <LLOQ and post-vaccination titer >=4*LLOQ or (2) Pre-dose titer >LLOQ and post-vaccination titer >=4*pre-dose 1 titer value. As specified in the protocol, data for this outcome measure was not collected and analyzed for Cohort 1: Ad26.COV2.S 2.5*10^10 vp and 1*10^10 vp participants.
Time Frame: 28 days after primary vaccination with Ad26.COV2.S (Day 29 of study VAC31518COV3001)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp)
Number analyzed (Participants) | 308
Percentage of participants | 8.8 [5.9 to 12.5]

8. Primary Outcome: Cohort 1: GMTs of Neutralizing Antibodies Against the Leading Variant of High Consequence or Concern (Delta Variant) 28 Days After Primary Vaccination With Ad26.COV2.S (5*10^10 vp Dose Level)
Description: GMTs of neutralizing antibodies against the leading variant of high consequence or concern (delta variant) 28 days after primary vaccination with Ad26.COV2.S (5*10^10 vp dose level) were reported. GMT against Delta variant was assessed by VNA. As specified in the protocol, data for this outcome measure was not collected and analyzed for Cohort 1: Ad26.COV2.S 2.5*10^10 vp and 1*10^10 vp participants. Lower limit of Quantification (LLOQ) was 65.
Time Frame: 28 days after primary vaccination with Ad26.COV2.S (Day 29 of study VAC31518COV3001)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp)
Number analyzed (Participants) | 311
Titer | NA [NA to NA] — Geometric mean and lower limit and upper limit of 95% CI could not be estimated as the lower and upper limit of 95% CI values were below the LLOQ (65).

9. Primary Outcome: Cohort 2: Percentage of Participants With Serological Response Against SARS-CoV-2 Original Strain, 14 Days After Ad26.COV2.S Booster Vaccination After Completing 2-dose Primary Vaccination With BNT162b2
Description: Percentage of participants with serological response against SARS-CoV-2 original strain, 14 days after Ad26.COV2.S booster vaccination after completing 2-dose primary vaccination with BNT162b2 were reported. A participant was considered a responder if at least one of the following conditions were satisfied: (1) If pre-booster 1 titer <LLOQ, then post-booster titer >=4*LLOQ or (2) If pre-booster 1 titer >LLOQ, then post-booster titer >=4*pre-booster value (titer).
Time Frame: 14 days after Ad26.COV2.S booster vaccination (i.e., On Day 15)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 297 | 294 | 88
Percentage of participants | 97.0 [94.3 to 98.6] | 90.5 [86.5 to 93.6] | 89.8 [81.5 to 95.2]

10. Primary Outcome: Cohort 2: GMTs of Neutralizing Antibodies Against SARS-CoV-2 Original Strain 14 Days After Ad26.COV2.S Booster Vaccination After Completing 2-dose Primary Vaccination With BNT162b2
Description: GMTs of neutralizing antibodies against SARS-CoV-2 original strain 14 days after Ad26.COV2.S booster vaccination after completing 2-dose primary vaccination with BNT162b2 were reported. GMT against original strain was assessed by VNA.
Time Frame: 14 days after Ad26.COV2.S booster vaccination (i.e., On Day 15)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 299 | 295 | 88
Titer | 4439 [4027 to 4893] | 3566 [3212 to 3958] | 3218 [2582 to 4010]

11. Primary Outcome: Cohort 2: Percentage of Participants With Serological Response Against SARS-CoV-2 Original Strain 2 Weeks to 2 Months After Completing 2-dose Primary Vaccination With BNT162b2 (Pfizer BNT162b2 External Samples)
Description: Percentage of participants with serological response against SARS-CoV-2 original strain 2 weeks to 2 months after completing 2-dose primary vaccination with BNT162b2 were planned to be reported. A participant was considered a responder if at least one of the following conditions were satisfied: (1) If pre-dose 1 titer <LLOQ, then post-vaccination titer >=4*LLOQ. (2) If pre-dose 1 titer >LLOQ, then post-vaccination titer >=4*pre-dose 1 value (titer).
Time Frame: 2 weeks to 2 months after primary vaccination with BNT162b2 (up to 1.5 months)
Population: Pre-dose data prior to primary vaccination with BNT162b2 was not collected and analyzed and thus the planned serological response data post-primary vaccination (BNT162b2) could not be estimated based on the protocol-defined serological response criteria.
Groups:
- Pfizer External Samples: Participants who received Pfizer vaccine BNT162b2 as primary vaccination were analyzed in this arm group.
Arm/Group | Pfizer External Samples
Number analyzed (Participants) | 0

12. Primary Outcome: Cohort 2: GMTs of Neutralizing Antibodies Against SARS-CoV-2 Original Strain 2 Weeks to 2 Months After Completing 2-dose Primary Vaccination With BNT162b2 (Pfizer BNT162b2 External Samples)
Description: GMTs of neutralizing antibodies against SARS-CoV-2 original strain 2 weeks to 2 months after completing 2-dose primary vaccination with BNT162b2 were reported. GMT against original strain was assessed by VNA.
Time Frame: 2 weeks to 2 months after primary vaccination with BNT162b2 (up to 1.5 months)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Pfizer External Samples
Number analyzed (Participants) | 309
Titer | 1281 [1086 to 1510]

13. Primary Outcome: Cohort 2: Percentage of Participants With Serological Response Against SARS-CoV-2 Delta Variant 14 Days After Booster Vaccination (5*10^10 vp Dose Level) After Completing 2-dose Primary Vaccination With BNT162b2
Description: Percentage of participants with serological response against SARS-CoV-2 leading variant of high consequence or concern (Delta) 14 days after booster vaccination (5*10^10 vp dose level) after completing 2-dose primary vaccination with BNT162b2 were reported. A participant was considered a responder if at least one of the following conditions was satisfied: (1) If pre-booster 1 titer <LLOQ, then post-booster titer >=4*LLOQ or (2) If pre-booster 1 titer >LLOQ, then post-booster titer >=4*pre-booster value (titer). As specified in the protocol, data for this outcome measure was not collected and analyzed for Cohort 2: Ad26.COV2.S 2.5*10^10 vp and 1*10^10 vp participants.
Time Frame: 14 days after Ad26.COV2.S booster vaccination (i.e., On Day 15)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Ad26.COV2.S (5*10^10 vp)
Number analyzed (Participants) | 297
Percentage of participants | 93.6 [90.2 to 96.1]

14. Primary Outcome: Cohort 2: GMTs of Neutralizing Antibodies Against the SARS-CoV-2 Leading Variant of High Consequence or Concern (Delta Variant) 14 Days After Booster Vaccination (5*10^10 vp Dose Level) After Completing 2-dose Primary Vaccination With BNT162b2
Description: Antibody GMTs of neutralizing antibodies against the SARS-CoV-2 leading variant of high consequence or concern (Delta variant) 14 days after booster vaccination after completing 2-dose primary vaccination with BNT162b2 were reported. GMT against delta variant was assessed by VNA. As specified in the protocol, data for this outcome measure was not collected and analyzed for Cohort 2: Ad26.COV2.S 2.5*10^10 vp and 1*10^10 vp participants.
Time Frame: 14 days after Ad26.COV2.S booster vaccination (i.e., On Day 15)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 2: Ad26.COV2.S (5*10^10 vp)
Number analyzed (Participants) | 299
Titer | 2318 [2049 to 2623]

15. Primary Outcome: Cohort 2: Percentage of Participants With Seropositive Response to Vaccination Against the SARS-CoV-2 Delta Variant 2 Weeks to 2 Months After Completing Primary Vaccination With 2-dose BNT162b2 (Pfizer BNT162b2 External Samples)
Description: Percentage of participants with seropositive response to vaccination against the SARS-CoV-2 leading variant of high consequence or concern (Delta) 2 weeks to 2 months after completing primary vaccination with 2-dose BNT162b2 were planned to be reported. A participant was considered a responder if one or both of the following conditions was satisfied: (1) Pre-dose titer <LLOQ and post-vaccination titer >=4*LLOQ. or (2) Pre-dose titer >LLOQ and post-vaccination titer >=4*pre-dose 1 titer value.
Time Frame: 2 weeks to 2 months after primary vaccination with BNT162b2 (up to 1.5 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pfizer External Samples
Number analyzed (Participants) | 309
Percentage of participants | 83.8 [79.2 to 87.7]

16. Primary Outcome: Cohort 2: GMTs of Neutralizing Antibodies Against the SARS-CoV-2 Delta Variant 2 Weeks to 2 Months After Completing 2-dose Primary Vaccination With BNT162b2 (Pfizer BNT162b2 External Samples)
Description: Antibody GMTs of neutralizing antibodies against the SARS-CoV-2 leading variant of high consequence or concern (Delta variant) 2 weeks to 2 months after completing 2-dose primary vaccination with BNT162b2 were reported. GMT against delta variant was assessed by VNA.
Time Frame: 2 weeks to 2 months after primary vaccination with BNT162b2 (up to 1.5 months)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Pfizer External Samples
Number analyzed (Participants) | 309
Titer | 502 [422 to 598]

17. Secondary Outcome: Cohorts 1 and 2: Number of Participants With Solicited Local Adverse Events (AEs) After Ad26.COV2.S Booster Vaccination
Description: Participants who received the booster dose were asked to note the occurrence of injection site pain, erythema, and swelling at the study vaccine injection site in e-Diary daily for 7 days post-booster vaccination (day of vaccination and the subsequent 7 days).
Time Frame: Up to 7 days after booster vaccination (Up to Day 8)
Population: Full analysis set (FAS) included all participants with a documented study vaccine administration (Ad26.COV2.S).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp) | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 330 | 326 | 116 | 326 | 328 | 106
Participants | 197 | 149 | 51 | 256 | 243 | 61

18. Secondary Outcome: Cohorts 1 and 2: Number of Participants With Solicited Systemic AEs After Ad26.COV2.S Booster Vaccination
Description: Participants recorded the temperature in the e-Diary in the evening of the day of vaccination, and then daily for the next 7 days approximately at the same time each day. If more than 1 measurement was made on any given day, the highest temperature of that day was recorded in the e-Diary. Fever was defined as endogenous elevation of body temperature >= 38.0 degree Celsius or >=100.4-degree Fahrenheit, as recorded in at least 1 measurement. Participants also noted the signs and symptoms in the e-Diary on a daily basis for 7 days post-booster vaccination (day of vaccination and the subsequent 7 days), if feasible, for the following events: fatigue, headache, nausea, myalgia.
Time Frame: Up to 7 days after booster vaccination (Up to Day 8)
Population: FAS included all participants with a documented study vaccine administration (Ad26.COV2.S).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp) | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 330 | 326 | 116 | 326 | 328 | 106
Participants | 188 | 160 | 60 | 267 | 234 | 67

19. Secondary Outcome: Cohorts 1 and 2: Number of Participants With Unsolicited AEs After Ad26.COV2.S Booster Vaccination
Description: Unsolicited AEs were all AEs for which the participant was not specifically questioned in the participant diary.
Time Frame: Up to 28 days after booster vaccination (Up to Day 29)
Population: FAS included all participants with a documented study vaccine administration (Ad26.COV2.S).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp) | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 330 | 326 | 116 | 326 | 328 | 106
Participants | 37 | 35 | 14 | 55 | 56 | 16

20. Secondary Outcome: Cohorts 1 and 2: Number of Participants With Serious Adverse Events (SAEs) After Ad26.COV2.S Booster Vaccination
Description: SAE is any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: From booster vaccination (Day 1) until 1 year post booster vaccination
Population: FAS included all participants with a documented study vaccine administration (Ad26.COV2.S).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp) | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 330 | 326 | 116 | 326 | 328 | 106
Participants | 11 | 7 | 2 | 9 | 4 | 2

21. Secondary Outcome: Cohorts 1 and 2: Number of Participants With Adverse Events of Special Interest (AESIs) After Ad26.COV2.S Booster Vaccination
Description: Number of participants with AESIs were reported. AESIs are significant AEs that are judged to be of special interest because of clinical importance, known or suspected class effects, or based on nonclinical signals.
Time Frame: From booster vaccination (Day 1) until 1 year post booster vaccination
Population: FAS included all participants with a documented study vaccine administration (Ad26.COV2.S).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp) | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 330 | 326 | 116 | 326 | 328 | 106
Participants | 2 | 5 | 0 | 1 | 0 | 0

22. Secondary Outcome: Cohort 1: Percentage of Participants With Serological Response Against SARS-CoV-2 Original Strain, Delta, and Beta Variant 14 Days After Ad26.COV2.S Booster Vaccination After Primary Vaccination With Ad26.COV2.S
Description: Percentage of participants with serological response against SARS-CoV-2 original strain, leading variant of high consequence or concern (delta variant), and other relevant variant of concern (beta variant) 14 days after Ad26.COV2.S booster vaccination after primary vaccination with Ad26.COV2.S were reported. A participant was considered a responder if at least one of the following conditions were satisfied: (1) If pre-booster 1 titer <LLOQ, then post-booster titer >=4*LLOQ or (2) If pre-booster 1 titer >LLOQ, then post-booster titer >=4*pre-booster value (titer).
Time Frame: 14 days after Ad26.COV2.S booster vaccination (i.e., On Day 15)
Population: Per protocol immunogenicity (PPI) population included all vaccinated participants for whom post-baseline immunogenicity data were available excluding participants with major protocol deviations expected to impact the immunogenicity outcomes. Here, N (Overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 298 | 297 | 93
Percentage of participants
  Original Strain | 63.4 [57.7 to 68.9] | 57.9 [52.1 to 63.6] | 64.5 [53.9 to 74.2]
  Delta Variant | 56.7 [50.9 to 62.4] | 49.2 [43.3 to 55.0] | 51.6 [41.0 to 62.1]
  Beta Variant | 40.9 [35.3 to 46.8] | 32.0 [26.7 to 37.6] | 18.3 [11.0 to 27.6]

23. Secondary Outcome: Cohort 1: Percentage of Participants With Serological Response Against SARS-CoV-2 Leading Variant of High Consequence or Concern (Omicron Variant) 14 Days After Ad26.COV2.S Booster Vaccination After Primary Vaccination With Ad26.COV2.S
Description: Percentage of participants with serological response against SARS-CoV-2 leading variant of high consequence or concern (omicron variant) 14 days after Ad26.COV2.S booster vaccination after primary vaccination with Ad26.COV2.S were reported.
Time Frame: 14 days after Ad26.COV2.S booster vaccination (i.e., On Day 15)
Population: PPI population included all vaccinated participants for whom post-baseline immunogenicity data were available excluding participants with major protocol deviations expected to impact the immunogenicity outcomes. Here, N (Overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 270 | 257 | 78
Percentage of participants | 9.6 [6.4 to 13.8] | 8.2 [5.1 to 12.2] | 6.4 [2.1 to 14.3]

24. Secondary Outcome: Cohort 1: GMTs of Neutralizing Antibodies Against the Original Strain, Delta and Beta Strain 14 Days After Ad26.COV2.S Booster Vaccination
Description: GMTs of neutralizing antibodies against the original strain, leading variant of high consequence or concern (delta variant), and other relevant variant of concern (beta variant) 14 days after Ad26.COV2.S booster vaccination were reported. GMT against original strain was assessed by VNA.
Time Frame: 14 days after Ad26.COV2.S booster vaccination (i.e., On Day 15)
Population: as for outcome 23
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 298 | 297 | 93
Titer
  Original Strain | 1130 [989 to 1291] | 915 [792 to 1058] | 734 [564 to 954]
  Delta Variant | 471 [411 to 539] | 391 [335 to 456] | 316 [244 to 409]
  Beta Variant | 274 [240 to 314] | 237 [205 to 275] | 156 [125 to 194]

25. Secondary Outcome: Cohort 1: GMTs of Neutralizing Antibodies Against the Leading Variant of High Consequence or Concern (Omicron Variant) 14 Days After Ad26.COV2.S Booster Vaccination
Description: GMTs of neutralizing antibodies against the leading variant of high consequence or concern (omicron variant) 14 days after Ad26.COV2.S booster vaccination were reported.
Time Frame: 14 days after Ad26.COV2.S booster vaccination (i.e., On Day 15)
Population: as for outcome 23
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 270 | 257 | 78
Titer | 69 [NA to 78] — Lower limit of 95% CI could not be estimated as it was below the LLOQ (66). | 71 [NA to 81] — Lower limit of 95% CI could not be estimated as it was below the LLOQ (66). | NA [NA to 69] — Geometric mean and lower limit of 95% CI could not be estimated as it was below the LLOQ (66).

26. Secondary Outcome: Cohort 1: Percentage of Participants With Serological Response Against SARS-CoV-2 Original Strain, Delta, and Beta Variant 28 Days After Ad26.COV2.S Booster Vaccination After Primary Vaccination With Ad26.COV2.S
Description: Percentage of participants with serological response against SARS-CoV-2 original strain, leading variant of high consequence or concern (delta variant), and other relevant variant of concern (beta variant) 28 days after Ad26.COV2.S booster vaccination after primary vaccination with Ad26.COV2.S were reported. A participant was considered a responder if at least one of the following conditions were satisfied: (1) If pre-booster 1 titer <LLOQ, then post-booster titer >=4*LLOQ or (2) If pre-booster 1 titer >LLOQ, then post-booster titer >=4*pre-booster value (titer).
Time Frame: 28 days after Ad26.COV2.S booster vaccination (i.e., On Day 29)
Population: PPI population included all vaccinated participants for whom post-baseline immunogenicity data were available excluding participants with major protocol deviations expected to impact the immunogenicity outcomes. Here, N (Overall number of participants analyzed) signifies participants with available data for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 32 | 33 | 24
Percentage of participants
  Original Strain | 68.8 [50.0 to 83.9] | 63.6 [45.1 to 79.6] | 75.0 [53.3 to 90.2]
  Delta Variant | 59.4 [40.6 to 76.3] | 36.4 [20.4 to 54.9] | 62.5 [40.6 to 81.2]
  Beta Variant | 40.6 [23.7 to 59.4] | 18.2 [7.0 to 35.5] | 29.2 [12.6 to 51.1]

27. Secondary Outcome: Cohort 1: Percentage of Participants With Serological Response Against SARS-CoV-2 Leading Variant of High Consequence or Concern (Omicron Variant) 28 Days After Ad26.COV2.S Booster Vaccination After Primary Vaccination With Ad26.COV2.S
Description: Percentage of participants with serological response against SARS-CoV-2 leading variant of high consequence or concern (omicron variant) 28 days after Ad26.COV2.S booster vaccination after primary vaccination with Ad26.COV2.S were reported.
Time Frame: 28 days after Ad26.COV2.S booster vaccination (i.e., On Day 29)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 32 | 29 | 23
Percentage of participants | 9.4 [2.0 to 25.0] | 6.9 [0.8 to 22.8] | 4.30 [0.1 to 21.9]

28. Secondary Outcome: Cohort 1: GMTs of Neutralizing Antibodies Against the Original Strain, Delta and Beta Strain 28 Days After Ad26.COV2.S Booster Vaccination
Description: GMTs of neutralizing antibodies against the original strain, leading variant of high consequence or concern (delta variant), and other relevant variant of concern (beta variant) 28 days after Ad26.COV2.S booster vaccination were reported. GMT was assessed by VNA.
Time Frame: 28 days after Ad26.COV2.S booster vaccination (i.e., On Day 29)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 32 | 33 | 24
Titer
  Original Strain | 993 [688 to 1434] | 893 [546 to 1459] | 887 [559 to 1408]
  Delta Variant | 455 [320 to 647] | 328 [197 to 545] | 333 [183 to 608]
  Beta Variant | 269 [188 to 384] | 201 [127 to 321] | 190 [116 to 311]

29. Secondary Outcome: Cohort 1: GMTs of Neutralizing Antibodies Against the Leading Variant of High Consequence or Concern (Omicron Variant) 28 Days After Ad26.COV2.S Booster Vaccination
Description: GMTs of neutralizing antibodies against the leading variant of high consequence or concern (omicron variant) 28 days after Ad26.COV2.S booster vaccination were reported.
Time Frame: 28 days after Ad26.COV2.S booster vaccination (i.e., On Day 29)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 32 | 29 | 23
Titer | 77 [NA to 108] — Lower limit of 95% CI could not be estimated as it was below the LLOQ (66). | NA [NA to 92] — Geometric mean and lower limit of 95% CI could not be estimated as it was below the LLOQ (66). | NA [NA to 85] — Geometric mean and lower limit of 95% CI could not be estimated as it was below the LLOQ (66).

30. Secondary Outcome: Cohort 1: Percentage of Participants With Antibodies Binding to SARS-CoV-2 Relevant Variants of Concern or Individual SARS-CoV-2 Proteins by Enzyme-linked Immunosorbent Assay (ELISA)
Description: Percentage of participants with antibodies binding to SARS-CoV-2 relevant variants of concern or individual SARS-CoV-2 Proteins by ELISA were planned to be reported.
Time Frame: 28 days after Ad26.COV2.S booster vaccination (i.e., On Day 29)
Population: PPI population was analyzed. Here, N (Overall number of participants analyzed) signifies participants with available data for this outcome measure and "0" in the number analyzed field signifies that no participants were available for the analysis because data of antibodies binding to SARS-CoV-2 relevant variants of concern was not collected and analyzed due to change in planned analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 32 | 29 | 23
Percentage of participants
  SARS-CoV-2 Relevant Variants of Concern: number analyzed (Participants) | 0 | 0 | 0
  Individual SARS-CoV-2 Proteins | 100.0 [89.1 to 100.0] | 96.6 [82.2 to 99.9] | 100.0 [85.2 to 100.0]

31. Secondary Outcome: Cohort 1: Number of Participants With Antibodies Binding to SARS-CoV-2 Relevant Variants of Concern or Individual SARS-CoV-2 Proteins by Meso Scale Discovery (MSD)
Description: Number of participants with antibodies binding to SARS-CoV-2 relevant variants of concern or individual SARS-CoV-2 Proteins by MSD were planned to be reported.
Time Frame: From booster vaccination (Day 1) until 1 year from booster vaccination
Population: Data for this outcome measure was not collected and analyzed due to change in planned analysis.
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 0 | 0 | 0

32. Secondary Outcome: Cohort 2: Percentage of Participants With Serological Response to Vaccination Against the Original Strain, Delta and Beta Variant 14 Days After Ad26.COV2.S Booster Vaccination After Primary Vaccination With BNT162b2
Description: Percentage of participants with serological response to vaccination against the original strain, leading variant of high consequence or concern (delta variant), and other relevant variant of concern (beta variant) 14 days after Ad26.COV2.S booster vaccination after primary vaccination with BNT162b2 were reported. A participant was considered a responder if at least one of the following conditions was satisfied: (1) If pre-booster 1 titer <LLOQ, then post-booster titer >=4*LLOQ or (2) If pre-booster 1 titer >LLOQ, then post-booster titer >=4*pre-booster value (titer).
Time Frame: 14 days after Ad26.COV2.S booster vaccination (i.e., On Day 15)
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 297 | 294 | 88
Percentage of participants
  Original Strain | 97.0 [94.3 to 98.6] | 90.5 [86.5 to 93.6] | 89.8 [81.5 to 95.2]
  Delta Variant | 93.6 [90.2 to 96.1] | 91.2 [87.3 to 94.1] | 86.4 [77.4 to 92.8]
  Beta Variant | 88.2 [84.0 to 91.7] | 82.7 [77.8 to 86.8] | 78.4 [68.4 to 86.5]

33. Secondary Outcome: Cohort 2: Percentage of Participants With Serological Response to Vaccination Against the Leading Variant of High Consequence or Concern (Omicron Variant) 14 Days After Ad26.COV2.S Booster Vaccination After Primary Vaccination With BNT162b2
Description: Percentage of participants with serological response to vaccination against the leading variant of high consequence or concern (omicron variant) 14 days after Ad26.COV2.S booster vaccination after primary vaccination with BNT162b2 was reported.
Time Frame: 14 days after Ad26.COV2.S booster vaccination (i.e., On Day 15)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 299 | 295 | 89
Percentage of participants | 72.5 [67.0 to 77.5] | 62.0 [56.2 to 67.6] | 56.2 [45.3 to 66.7]

34. Secondary Outcome: Cohort 2: Antibody GMTs of Neutralizing Antibodies Against the Original Strain, Delta and Beta Variant 14 Days After Ad26.COV2.S Booster Vaccination After Completing Primary Vaccination With BNT162b2
Description: Antibody GMTs of neutralizing antibodies against the original strain, leading variant of high consequence or concern (delta variant), and other relevant variant of concern (beta variant) 14 days after Ad26.COV2.S booster vaccination after completing primary vaccination with BNT162b2 were reported.
Time Frame: 14 days after Ad26.COV2.S booster vaccination (i.e., On Day 15)
Population: as for outcome 23
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 299 | 295 | 88
Titer
  Original Strain | 4439 [4027 to 4893] | 3566 [3212 to 3958] | 3218 [2582 to 4010]
  Delta Variant | 2318 [2049 to 2623] | 1872 [1646 to 2129] | 1761 [1372 to 2261]
  Beta Variant | 1649 [1432 to 1900] | 1310 [1135 to 1511] | 1055 [787 to 1412]

35. Secondary Outcome: Cohort 2: Antibody GMTs of Neutralizing Antibodies Against the Leading Variant of High Consequence or Concern (Omicron Variant) 14 Days After Ad26.COV2.S Booster Vaccination After Completing Primary Vaccination With BNT162b2
Description: Antibody GMTs of neutralizing antibodies against the leading variant of high consequence or concern (omicron variant) 14 days after Ad26.COV2.S booster vaccination after completing primary vaccination with BNT162b2 were reported.
Time Frame: 14 days after Ad26.COV2.S booster vaccination (i.e., On Day 15)
Population: as for outcome 23
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 299 | 295 | 89
Titer | 509 [440 to 590] | 386 [327 to 455] | 336 [252 to 449]

36. Secondary Outcome: Cohort 2: Percentage of Participants With Serological Response to Vaccination Against the Original Strain, Delta and Beta Variant 28 Days After Ad26.COV2.S Booster Vaccination After Primary Vaccination With BNT162b2
Description: Percentage of participants with serological response to vaccination against the original strain, leading variant of high consequence or concern (delta variant), and other relevant variant of concern (Beta variant) 28 days after Ad26.COV2.S booster vaccination after primary vaccination with BNT162b2 were reported. A participant was considered a responder if at least one of the following conditions was satisfied: (1) If pre-booster 1 titer <LLOQ, then post-booster titer >=4*LLOQ or (2) If pre-booster 1 titer >LLOQ, then post-booster titer >=4*pre-booster value (titer).
Time Frame: 28 days after Ad26.COV2.S booster vaccination (i.e., On Day 29)
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 35 | 33 | 23
Percentage of participants
  Original Strain | 100.0 [90.0 to 100.0] | 97.0 [84.2 to 99.9] | 95.7 [78.1 to 99.9]
  Delta Variant | 97.1 [85.1 to 99.9] | 97.0 [84.2 to 99.9] | 87.0 [66.4 to 97.2]
  Beta Variant | 94.3 [80.8 to 99.3] | 78.8 [61.1 to 91.0] | 82.6 [61.2 to 95.0]

37. Secondary Outcome: Cohort 2: Percentage of Participants With Serological Response to Vaccination Against the Leading Variant of High Consequence or Concern (Omicron Variant) 28 Days After Ad26.COV2.S Booster Vaccination After Primary Vaccination With BNT162b2
Description: Percentage of participants with serological response to vaccination against the leading variant of high consequence or concern (omicron variant) 28 days after Ad26.COV2.S booster vaccination after primary vaccination with BNT162b were reported.
Time Frame: 28 days after Ad26.COV2.S booster vaccination (i.e., On Day 29)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 35 | 33 | 23
Percentage of participants | 77.1 [59.9 to 89.6] | 57.6 [39.2 to 74.5] | 69.6 [47.1 to 86.8]

38. Secondary Outcome: Cohort 2: GMTs of Neutralizing Antibodies Against the Original Strain, Delta and Beta Strain 28 Days After Ad26.COV2.S Booster Vaccination After Completing Primary Vaccination With BNT162b2
Description: GMTs of neutralizing antibodies against the original strain, leading variant of high consequence or concern (delta variant), and other relevant variant of concern (beta variant) 28 days after Ad26.COV2.S booster vaccination after completing primary vaccination with BNT162b2 were reported.
Time Frame: 28 days after Ad26.COV2.S booster vaccination (i.e., On Day 29)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 35 | 33 | 23
Titer
  Original Strain | 6221 [4905 to 7890] | 4808 [3496 to 6612] | 4410 [3067 to 6341]
  Delta Variant | 3414 [2358 to 4944] | 2348 [1584 to 3480] | 1803 [1138 to 2855]
  Beta Variant | 2144 [1426 to 3226] | 1614 [1031 to 2529] | 1116 [579 to 2152]

39. Secondary Outcome: Cohort 2: GMTs of Neutralizing Antibodies Against the Leading Variant of High Consequence or Concern (Omicron Variant) 28 Days After Ad26.COV2.S Booster Vaccination After Completing Primary Vaccination With BNT162b2
Description: GMTs of neutralizing antibodies against the leading variant of high consequence or concern (omicron variant) 28 days after Ad26.COV2.S booster vaccination after completing primary vaccination with BNT162b2 were reported.
Time Frame: 28 days after Ad26.COV2.S booster vaccination (i.e., On Day 29)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 35 | 33 | 23
Titer | 752 [496 to 1140] | 452 [282 to 724] | 391 [211 to 725]

40. Secondary Outcome: Cohort 2: Percentage of Participants With Antibodies Binding to SARS-CoV-2 Relevant Variants of Concern or Individual SARS-CoV- 2 Proteins by ELISA
Description: Percentage of participants with antibodies binding to SARS-CoV-2 relevant variants of concern or individual SARS-CoV- 2 proteins by ELISA were planned to be reported.
Time Frame: 28 days after Ad26.COV2.S booster vaccination (i.e., On Day 29)
Population: as for outcome 30
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 35 | 33 | 23
Percentage of participants
  SARS-CoV-2 Relevant Variants of Concern: number analyzed (Participants) | 0 | 0 | 0
  Individual SARS-CoV-2 Proteins | 100.0 [90.0 to 100.0] | 100.0 [89.4 to 100.0] | 100.0 [85.2 to 100.0]

41. Secondary Outcome: Cohort 2: Number of Participants With Antibodies Binding to SARS-CoV-2 Relevant Variants of Concern or Individual SARS-CoV- 2 Proteins by MSD
Description: Number of participants with antibodies binding to SARS-CoV-2 relevant variants of concern or individual SARS-CoV- 2 proteins by MSD were planned to be reported.
Time Frame: From booster vaccination (Day 1) until 1 year from booster vaccination
Population: Data for this outcome measure was not collected and analyzed due to change in planned analysis.
Arm/Group | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 0 | 0 | 0

42. Secondary Outcome: Cohorts 1 and 2: Number of Participants With Antibodies Binding to the SARS-CoV-2 Nucleocapsid (N) Protein at Day 1 as Assessed by N-Serology
Description: Number of participants with antibodies binding to the SARS-CoV-2 nucleocapsid (N) protein at Day 1 as assessed by N-serology were planned to be reported.
Time Frame: Day 1
Population: Data for this outcome measure was not collected and analyzed due to change in planned analysis.
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp) | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From booster vaccination (Day 1) until 1 year post booster vaccination
Description: FAS included all participants with a documented study vaccine administration (Ad26.COV2.S).
Arm/Group | Cohort 1: Ad26.COV2.S (5*10^10 vp) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) | Cohort 1: Ad26.COV2.S (1*10^10 vp) | Cohort 2: Ad26.COV2.S (5*10^10 vp) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) | Cohort 2: Ad26.COV2.S (1*10^10 vp)
All-Cause Mortality (participants affected / at risk) | 1/330 | 1/326 | 0/116 | 0/326 | 0/328 | 0/106
Serious Adverse Events (participants affected / at risk) | 11/330 | 7/326 | 2/116 | 9/326 | 4/328 | 2/106
Other Adverse Events (participants affected / at risk) | 239/330 | 201/326 | 75/116 | 294/326 | 271/328 | 77/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Ad26.COV2.S (5*10^10 vp) (N=330) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) (N=326) | Cohort 1: Ad26.COV2.S (1*10^10 vp) (N=116) | Cohort 2: Ad26.COV2.S (5*10^10 vp) (N=326) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) (N=328) | Cohort 2: Ad26.COV2.S (1*10^10 vp) (N=106)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Systemic Inflammatory Response Syndrome (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Biliary Obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Endometritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Posterior Tibial Tendon Dysfunction (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rib Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Ovarian Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Thoracic Outlet Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bipolar Disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Spinal Fusion Surgery (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Spinal Laminectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Giant Cell Arteritis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Ad26.COV2.S (5*10^10 vp) (N=330) | Cohort 1: Ad26.COV2.S (2.5*10^10 vp) (N=326) | Cohort 1: Ad26.COV2.S (1*10^10 vp) (N=116) | Cohort 2: Ad26.COV2.S (5*10^10 vp) (N=326) | Cohort 2: Ad26.COV2.S (2.5*10^10 vp) (N=328) | Cohort 2: Ad26.COV2.S (1*10^10 vp) (N=106)
Nausea (Gastrointestinal disorders) | 49 | 42 | 11 | 102 | 75 | 12
Fatigue (General disorders) | 154 | 119 | 46 | 234 | 194 | 53
Malaise (General disorders) | 3 | 4 | 3 | 1 | 0 | 1
Pyrexia (General disorders) | 4 | 6 | 1 | 32 | 19 | 1
Vaccination Site Erythema (General disorders) | 4 | 3 | 1 | 9 | 10 | 1
Vaccination Site Pain (General disorders) | 196 | 149 | 50 | 256 | 242 | 61
Vaccination Site Swelling (General disorders) | 4 | 2 | 0 | 5 | 8 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 3 | 1 | 8 | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 110 | 87 | 28 | 198 | 168 | 35
Headache (Nervous system disorders) | 110 | 91 | 34 | 214 | 154 | 43
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 3 | 2 | 3 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 4 | 4 | 4 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 3 | 2 | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. Expedited reviews will be arranged for abstracts, poster presentations, or other materials. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT04999111/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT04999111/SAP_002.pdf